CLINICAL TRIAL: NCT04749043
Title: Virtual Reality Compared to Nitrous Oxide for Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brendan Carvalho (Other)
Responsible Party: Sponsor-Investigator, Brendan Carvalho, Chief, Division of Obstetric Anesthesia, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 59344
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Labor Pain
Keywords: Virtual Reality
MeSH Terms: conditions — Labor Pain | interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: Comparing VR to an "active control" of nitrous oxide as a current standard of care for non-epidural analgesic in a crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality then Nitrous Oxide (Active Comparator): 30 minute exposure to virtual reality, 5 minute washout period, then 30 minute exposure to nitrous oxide
  Interventions: Device: Oculus Quest 2 Virtual Reality Device; Drug: Nitrous oxide
- Nitrous Oxide then Virtual Reality (Active Comparator): 30 minute exposure to nitrous oxide, 5 minute washout period, then 30 minute exposure to virtual reality
  Interventions: Device: Oculus Quest 2 Virtual Reality Device; Drug: Nitrous oxide

INTERVENTIONS:
Device: Oculus Quest 2 Virtual Reality Device — 30 min VR experience exposure for labor analgesia. VR experiences include swimming in the ocean, walking through forests, engaging in 3D puzzles, exploring virtual lands, or interacting with musical objects
Drug: Nitrous oxide — 30 min exposure for labor analgesia

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headsets) are non-inferior to conventional therapy (nitrous oxide) for addressing maternal needs during labor who desire non-epidural pain relief.

DETAILED DESCRIPTION:
The investigators will use a commercially available consumer-grade virtual reality (VR) device and nitrous oxide, a standard of care therapy for laboring women desiring non-epidural analgesic, to determine satisfaction with pain relief with each therapy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy at >34 weeks
* Regular uterine contractions
* Pain > 2/10
* English speaking

Exclusion Criteria:

* BMI > 40
* Preeclampsia with severe features
* Use of IV analgesics during labor
* Diabetes requiring insulin therapy
* Claustrophobia
* History of epilepsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 70 minutes
  Patient satisfaction with pain relief on a scale of 0-10

SECONDARY OUTCOMES:
Pain score | 70 minutes
  Pain level on a scale of 0-10
Anxiety | 70 minutes
  Anxiety level on a scale of 0-10
Nausea | 70 minutes
  Nausea level on a scale of 0-10
Dizzy | 70 minutes
  Dizziness level on a scale of 0-10
Effectiveness | 70 minutes
  Effectiveness of device in relieving pain on a scale of 0-10
Cope with Pain | 70 minutes
  Ability to cope with pain on a scale of 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No